CLINICAL TRIAL: NCT05304806
Title: Effective Volemia in Older Adults With Orthostatic Hypotension, Feasibility Study
Brief Title: Effective Volemia in Older Adults With Orthostatic Hypotension
Acronym: EVO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220078; 2021-A03112-39 (Other: IDRCB)
Record Dates: First submitted 2022-02-09; First posted 2022-03-31 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Orthostatic Hypotension
Keywords: older; orthostatic hypotension; volemia; clinical sonography
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical and biological assessments of volemia are challenging in older patients as they are more likely to present non-typical signs. Point of care ultrasonography (POCUS) using heart and lung exploration is a relevant tool to assess volemia in adults with little data in older adults.

The primary objective of the study is to evaluate feasibility of positional POCUS in aging patients.

The secondary objectives are to assess the variability of measurements between decubitus and sitting position.

DETAILED DESCRIPTION:
This is a monocentric study. Twenty patients will be enrolled, aged of 70 years and older. POCUS parameters, duration of procedure and measurements will be recorded for each patients.

ELIGIBILITY:
Inclusion Criteria:

* 70 years and older
* Orthostatic hypotension or venous insufficiency
* Affiliated to a social security or beneficiary

Exclusion Criteria:

* Refusal to participation to the study
* Cognitive disorder
* Unable to keep sitting posture for up to 30 minutes
* Foreign patients under french AME scheme

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients older than 70 years, orthostatic hypotension
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-10-21 (Actual)

PRIMARY OUTCOMES:
Duration of recording during positional echography | 3 months
  Feasibility of positional echography assessed by
  - Duration of recording (minutes)
Feasibility of positional echography | 3 months
  Feasibility of positional echography assessed by
  - Number of good quality imaging (out of 5 pre specified views : parasternal long axis view, parasternal short axis view, apical views 4 and 5 chamber, subxiphoid view, inferior vena cava view)

SECONDARY OUTCOMES:
Cardiac ultra sound parameters: left ventricle diastolic diameter | 3 months
  - Left ventricle diastolic diameter mm/m2
Cardiac ultra sound parameters: left ventricle ejection fraction | 3 months
  - Left ventricle ejection fraction (%)
Cardiac ultra sound parameters: E and A waves velocity | 3 months
  - E and A waves velocity (cm/sec) (mitral Doppler)
Cardiac ultra sound parameters: Inferior vena cava size and compliance | 3 months
  - Inferior vena cava size (mm) and compliance (%)
Cardiac ultra sound parameters: left atrial size | 3 months
  - Left atrial size (cm2)

CONTACTS AND LOCATIONS:
Overall Officials: Marion Pepin, MD, PhD, Principal Investigator — Geriatric medecine department, Ambroise Paré hospital, APHP
Locations (1):
- Geriatric medecine department, Ambroise Paré hospital, APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No